CLINICAL TRIAL: NCT01318018
Title: Bilateral Bispectral Index Monitoring During and After Electroconvulsive Therapy Compared With Magnetic Seizure Therapy for Treatment-resistant Depression
Brief Title: Investigation on the Value of Bilateral Index (BIS) Monitoring for Magnetic Seizure Versus Electroconvulsive Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Martin Soehle, Consultant, University Hospital, Bonn
Other Study IDs: KTB
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2017-12

CONDITIONS: Depression
Keywords: depression; bispectral index; electroconvulsive therapy; magnetic seizure therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Magnetic Seizure Therapy Group: Patients receiving magnetic seizure therapy for depression
- Electroconvulsive Therapy Group: Patients receiving electroconvulsive therapy for depression

SUMMARY:
Electroconvulsive therapy (ECT) has been shown to be an effective treatment for patients suffering from depression, who do not respond to medical treatment. However it is often dismissed by patients, who feel uncomfortably about the application of electric shocks to their heads. In 2000, magnetic seizure therapy (MST) has been introduced which uses magnetism instead of electricity to evoke convulsions. MST seems to be as effective as ECT in terms of its antidepressant potency but may be associated with less severe cognitive side effects.

Control of anaesthesia during seizure therapy is demanding since light anesthesia might be associated with awareness, whereas deep anesthesia impedes the antidepressant effect of the convulsion. Therefore, Bispectral index (BIS) monitoring is frequently used to tailor anaesthesia for ECT, however little is known about BIS following MST.

The investigators hypothesize that in comparing MST with ECT, (a) patients show a faster increase in BIS and that (b)less left-right differences occur in BIS.

ELIGIBILITY:
Inclusion Criteria:

* depression

Exclusion Criteria:

* age < 18 years old
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from depression
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soehle, MD, PhD, Principal Investigator — Dept of Anaesthesiology and Intensive Care Medicine
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine & Dept. of Psychiatry and Psychotherapy, University of Bonn Hospital, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soehle M, Kayser S, Ellerkmann RK, Schlaepfer TE. Bilateral bispectral index monitoring during and after electroconvulsive therapy compared with magnetic seizure therapy for treatment-resistant depression. Br J Anaesth. 2014 Apr;112(4):695-702. doi: 10.1093/bja/aet410. Epub 2013 Dec 3. PMID 24305645
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnetic Seizure Therapy Group: Patients receiving magnetic seizure therapy for depression completed
Period: Overall Study
Arm/Group | Magnetic Seizure Therapy Group | Electroconvulsive Therapy Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnetic Seizure Therapy Group | Electroconvulsive Therapy Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14) | 55 (12) | 50 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time
Description: recovery time from seizure induction to eye opening / restoration of breathing
Time Frame: same day
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Magnetic Seizure Therapy Group: Patients receiving magnetic seizure therapy for depression recovery time
- Electroconvulsive Therapy Group: Patients receiving electroconvulsive therapy for depression recovery time
Arm/Group | Magnetic Seizure Therapy Group | Electroconvulsive Therapy Group
Number analyzed (Participants) | 10 | 10
minutes | 3.0 (1.0) | 6.7 (1.3)

ADVERSE EVENTS:
Groups:
- Magnetic Seizure Therapy Group: Patients receiving magnetic seizure therapy for depression: None
- Electroconvulsive Therapy Group: Patients receiving electroconvulsive therapy for depression: None
Arm/Group | Magnetic Seizure Therapy Group | Electroconvulsive Therapy Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes